CLINICAL TRIAL: NCT04080401
Title: Effectiveness of a Novel Gaming System on Post-operative Rehabilitation Outcomes After Total Knee Arthroplasty: A Pilot Study
Brief Title: Effectiveness of a Novel Gaming System on Post-operative Rehabilitation Outcomes After Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Ng Teng Fong Healthcare Innovation Programme (Unknown); Nanyang Technological University- UBC Research Centre in Active Living for the Elderly (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017/00229
Record Dates: First submitted 2019-08-14; First posted 2019-09-06 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Arthroplasty, Replacement; Physical Therapy
Keywords: Rehabilitation; Gaming; Exercise; Knee Arthroplasty
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fun-Knee Mobile Application (Experimental): Participants will use a mobile application paired to a knee sleeve with embedded inclinometer sensors. The sensor system will compute knee movement, and feed towards game-based rehabilitation exercises for Total Knee Arthroplasty rehabilitation. game-based and supported on mobile device running on Android or Inter-network Operating System platforms. The mobile apps is able to capture the angle and position data from the two inclinometers on smart knee sleeve.
  Interventions: Device: Game-based rehabilitation exercise
- Conventional Exercise Brochures (Active Comparator): Participants will be guided to do their Total Knee Arthroplasty rehabilitation exercises using conventional, paper-based exercise brochures.
  Interventions: Other: Conventional brochures of rehabilitation exercise

INTERVENTIONS:
Device: Game-based rehabilitation exercise — 4 games (exercises) on operated limb, for 3 sessions daily, until outpatient physiotherapy review visit.
  Arms: Fun-Knee Mobile Application
Other: Conventional brochures of rehabilitation exercise — 4 exercises on operated limb, 30 reps each, for 3 sessions daily, until outpatient physiotherapy review visit.
  Arms: Conventional Exercise Brochures

SUMMARY:
This study aims to evaluate the effectiveness of a novel, game-based rehabilitation system, consisting a sensor-equipped knee sleeve and a mobile application, on rehabilitation outcomes after Total Knee Arthroplasty (TKA) surgery, when compared to conventional rehabilitation; where patients learn and perform rehabilitative exercises using printed brochures.

DETAILED DESCRIPTION:
This is a randomized controlled trial investigating the effectiveness of a novel, game-based rehabilitation system, consisting a sensor-equipped knee sleeve and a mobile application, on rehabilitation outcomes after Total Knee Arthroplasty (TKA).

All patients receiving TKA will be screened for eligibility. Patients who meet inclusion criteria and provide informed consent will be allocated to either intervention or control group using block randomization. A study team member blinded to subject characteristics will allocate subjects to either group.

Subjects in the intervention group will be guided to do their post-TKA rehabilitation exercises using the investigator's game-based system, which includes the wearable sensor device and mobile application games. Subjects in the control group will be guided to do their post-TKA rehabilitation exercises using conventional, paper-based exercise brochures.

From post-operative day 1, all subjects who are medically fit for physiotherapy will receive 2 sessions of physiotherapy, daily; for at least the first 3 post-operative days. The first session consists of individualized physiotherapy that includes bed exercises and ambulation training. In the second session of physiotherapy, subjects will perform their bed exercises using the game-based system or paper-based exercise brochures. Upon discharge, subjects in the intervention group will continue home-based rehabilitation exercises using the game-based system, while those in the control group continue to use the exercise brochures.

ELIGIBILITY:
Inclusion Criteria:

* First, elective, unilateral TKA operation completed in Tan Tock Seng Hospital
* At least two days of inpatient stay
* Discharge to own or carer's home
* Adults >50 years old
* Able to understand and follow instructions consistently

Exclusion Criteria:

* Post-operative infections or wound complications
* Cognitive impairment
* Sensitive/ broken, Irritable skin around operative knee
* Previous TKA on same or opposite knee
* Pregnant women
* Pre-existing skin conditions e.g. eczema
* Poor wound status e.g. poor wound closure or condition

Min Age: 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Difference in pain score between hospital discharge and first outpatient physiotherapy review (within 3 weeks post-operation)
  Visual analogue scale (0-10) for participant-reported pain intensity. Maximum score (10) for worst pain, minimum score (0) for no pain.
Knee flexion range of motion | Difference in angle between hospital discharge and first outpatient physiotherapy review (within 3 weeks post-operation)
  Passive range of knee bending motion measured by handheld goniometry (ranging from -15 to 150 degrees), measuring angle formed by between femur and fibula.
Knee extension range of motion | Difference in angle between hospital discharge and first outpatient physiotherapy review (within 3 weeks post-operation)
  Passive range of knee straightening measured by handheld goniometry (ranging from -30 to 20 degrees), measuring angle formed by between femur and fibula.
Ambulation status | At hospital discharge, at outpatient review (2-3 weeks post-operation), at outpatient discharge or 3 months post-operation
  Use of gait aid, assistance during walking in the home or community

CONTACTS AND LOCATIONS:
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No